CLINICAL TRIAL: NCT07010913
Title: Erectile Dysfunction Progression After Coronary Angiography: Is Residual SYNTAX Score a Predictive Marker
Brief Title: Erectile Dysfunction Progression After Percutaneous Coronary Angiography: Is Residual SYNTAX Score a Predictive Marker
Status: Active, not recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Timucin Sipal, assistant Professor/ Lecturer, Kırıkkale University
Other Study IDs: 2025.01.13
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Coronary Arterial Disease (CAD); Erectile Dysfunction
Keywords: syntax score; residual syntax score; erectile disfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residual Syntax score more than 20%
- Residual Syntax score less than and equal 20%

SUMMARY:
Participant Information Sheet Dear Participant,

Investigators would like to invite participants to participate in a research study and explain what it involves. Please take a few moments to read the following information carefully. If you have any questions, feel free to ask us at any time.

What is this study about? This study aims to understand how coronary angiography (a heart procedure you've recently had) may affect erectile function over time. Investigators are especially interested in whether the degree of blockage in participants' heart vessels and how well participants were treated during the procedure affect erectile health.

What will participants be asked to do?

If participants agree to take part:

Investigators will ask participants to answer a short questionnaire with five questions about their erectile function. This will happen once while participants recover in the hospital and again 6 months later.

Each question is rated on a simple scale from 0 to 5.

Investigators will also collect some medical information, such as your age, weight, height, blood test results, details about your heart condition, other health problems, and the medications participants are taking.

All information will be kept confidential and used only for scientific purposes. Participants' identities will not be revealed in any part of the study.

Do participants have to take part? No. Participation is completely voluntary. Participants can choose not to take part, and you can also stop at any time without giving a reason. Participants' decisions will not affect their medical care in any way.

Will there be any extra tests or costs? No. This study does not involve extra tests beyond regular medical care, such as blood tests or heart monitoring, and participation is free.

How long will the study last? The study will last approximately one year. Once it's completed, participants are welcome to ask for the results from our institution.

Who is conducting the study?

The study is being conducted by:

Assist Prof Dr. Timucin Sipal (Urology Department)

Assist Prof Dr. Caglar Alp (Cardiology Department)

You can contact them anytime using the phone number we have provided.

What happens next? If participants are happy to participate, please sign the attached consent form.

Sincerely, The Research Team

ELIGIBILITY:
Inclusion Criteria:

* Having a First heart attack

Exclusion Criteria:

* History of previous coronary intervention
* Neurological condition
* Previous pelvic surgery
* Aged less than 20 and more than 70 years
* Having an additional heart attack during the follow-up period
* Excluding from the study
* Having no sexual life

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male erectile disfunction study
Study Population: Male participants who have a heart attack and undergo percutaneous coronary intervention in our institutions and survive the event.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Erectile functioning changes following percutaneous coronary intervention from baseline through 6 months | from February 2025 to September 2025
  Participants' answers will decrease or increase from the baseline score of 0 to 25 on the IIEF questionnaires following percutaneous coronary intervention after a heart attack.

CONTACTS AND LOCATIONS:
Locations (1):
- kirikkale Un'versity medical faculty, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: approximately at the end of August 2025